CLINICAL TRIAL: NCT04374058
Title: Reduced Frequency Hemodialysis in Prevalent Patients Due to the Coronavirus Disease
Brief Title: Less Frequency Hemodialysis and COVID-19
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Dialisis Madariaga (Other)
Responsible Party: Sponsor
Other Study IDs: coronavirus
Record Dates: First submitted 2020-05-01; First posted 2020-05-05 (Actual); Last update posted 2020-05-05 (Actual); Status verified 2020-05

CONDITIONS: End Stage Renal Disease
Keywords: Covid-19; Dialysis; less frequency hemodialysis; Ultrafiltration rate; Anemia; Nutrition
MeSH Terms: conditions — Kidney Failure, Chronic; COVID-19; Anemia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Two Times: The treatment group consists of selected patients that, based on their mean ultrafiltration rate, are switched from thrice-weekly to twice-weekly hemodialysis sessions
  Interventions: Other: less-frequency hemodialysis
- Three times: Usual thrice-weekly hemodialysis schedule
  Interventions: Other: less-frequency hemodialysis

INTERVENTIONS:
Other: less-frequency hemodialysis — Patients of treatment group would be evaluated quarterly

SUMMARY:
Facing the unusual situation imposed by the coronavirus disease, the aim of this study is to evaluate the risk and effects of less frequent hemodialysis on prevalent patients

DETAILED DESCRIPTION:
The novel coronavirus disease (COVID-19), also known as COVID-19 (and SARS-Cov2) by the World Health Organization, is a rapidly evolving pandemic. The outbreak is expected to infect a large portion of the world population, and a case fatality rate of 1-3% represents a significant mortality and healthcare burden. In common with other viral diseases, mortality is higher in elderly patients with high comorbidity.

The impressive figures of transmission in different communities underline the need for reorganization of efforts to limit contagion, particularly in crowded settings. Hemodialysis centres represents a specific setting in which many patients are repeatedly treated in the same area at the same time.

Dialysis patients constitute a susceptible population because of their older age, high comorbidity burden and their less efficient immune system. Therefore, they are more prone to develop severe infectious diseases than the general population.. Moreover, if infected, the requirements of specialized resources and staff is further complicated by requirements for isolation, control and prevention, putting healthcare systems under additional strain. Therefore, all measures to slow and to control unmanageably high incidence rates must be taken very seriously.

The routine treatment usually requires three dialysis sessions per week Further, some patients must travel long distances to the dialysis centre. One option to reduce the higher risk of these patients is to reduce the frequency of dialysis sessions.However, the potential benefits of reduced risk may be associated with higher interdialytic weight gain and inadequate dialysis, Two factors that increase the risk of mortality. Furthermore, the impact of reduced frequency on Anemia and Nutrition have not been extensively studied.

ELIGIBILITY:
Inclusion Criteria:

* More than 30 days of Chronic ambulatory in-center hemodialysis

Exclusion Criteria:

* More than three sessions a week
* amputated lower limbs

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The entire population of our satellite hemodialysis center, except those that meet the exclusion criteria, would be followed by one year
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2020-03-20 (Actual); Primary Completion 2021-03 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Mortality | From date of beginning of the study until the date of death assessed up to 52 weeks
  Time to all-cause and cardiovascular death

SECONDARY OUTCOMES:
Anemia, Nutrition, Adequation of dialysis, total ultrafiltration, ultrafiltration rate, | From date of beginning of the study assessed up to 52 weeks
  Time variation of the biological parameters mentioned in the title. Repeated measurements of laboratory variables will be averaged into patient quarterly means to minimize measurement variability.
Hospitalization | From date of beginning of the study until the date of first hospitalization assessed up to 52 weeks
  Time to first hospitalization of any cause
Vascular Access | From date of beginning of the study until the date of first intervention assessed up to 52 weeks
  Time to first endovascular or quirurgical intervention of the vascular access utilized at the start of the study

CONTACTS AND LOCATIONS:
Overall Officials: Esteban L Siga, MD, Principal Investigator — Dialisis Madariaga
Locations (1):
- Dialisis Madariaga, General Juan Madariaga, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: Undecided